CLINICAL TRIAL: NCT07001722
Title: Development and Implementation of an Online Psychological Support Program for Tobacco Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Ege University Scientific Research Projects Coordination (Unknown)
Responsible Party: Principal Investigator, Inci Derya YUCEL, Dr. Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-1.1T/38; 28432 (Other Grant/Funding Number: Ege University Office of Scientific Research Projects)
Record Dates: First submitted 2025-05-18; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Tobacco Addiction
Keywords: TUBSIS; tobacco use; mindfulness; web-based psychoeducation; Health Action Process Approach
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: The intervention is designed as a psychoeducational support remotely for tobacco user adult individuals. The control group had no intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TÜBSİS Web-based Psycho-education Programme (Experimental): The intervention group had the TÜBSİS Program, which consists of a total of 8 modules lasting 1 month, is supported by the integration of two different frameworks: Mindfulness Approach and HAPA Health Action Approach. While the progress process in the TÜBSİS Program was created with the HAPA Model, the module contents of it were created within the framework of the Mindfulness Approach. Each participant receives reminder emails during this asynchronous and distance learning process and can open each new module at least 3 days later.
  Participants in the intervention (as well as control group) were asked about sociodemographic and tobacco use characteristics at baseline. Health Action Process Approach (HAPA) Model Change Question Form, Warwick Edinburgh Mental Well-Being Scale, Fagerström Nicotine Dependence Test and Informed Consent Form were administered to the intervention group at the beginning, in the middle and at the end of the intervention study.
  Interventions: Other: TÜBSİS Web-based Psycho-education Programme
- Control Group (without intervention) (No Intervention): Participants in the control (as well as intervention group) were asked about sociodemographic and tobacco use characteristics at baseline. Health Action Process Approach (HAPA) Model Change Question Form, Warwick Edinburgh Mental Well-Being Scale, Fagerström Nicotine Dependence Test and Informed Consent Form were administered to the intervention group at the beginning, in the middle and at the end of the control study (during one month).

INTERVENTIONS:
Other: TÜBSİS Web-based Psycho-education Programme — The theoretical infrastructure of the TÜBSİS Program, which consists of a total of 8 modules lasting 1 month, is supported by the integration of two different frameworks: Mindfulness Approach and HAPA Health Action Approach. While the progress process in the TÜBSİS Program was created with the HAPA Model, the module contents of it were created within the framework of the Mindfulness Approach. Each participant receives reminder emails during this asynchronous and distance learning process and can open each new module at least 3 days later. Participants in the intervention (as well as control group) were asked about sociodemographic and tobacco use characteristics at baseline. Health Action Process Approach (HAPA) Model Change Question Form, Warwick Edinburgh Mental Well-Being Scale, Fagerström Nicotine Dependence Test and Informed Consent Form were administered to the intervention group at the beginning, in the middle and at the end of the intervention study.
  Arms: TÜBSİS Web-based Psycho-education Programme

SUMMARY:
Introduction: Tobacco use is the most prevalent and preventable public health problem in the world, responsible for 8 million deaths worldwide annually.

Objective: The aim of this study was to develop and implement a remote, asynchronous, eight-module psychoeducation programme (Tobacco Addiction Support System (TÜBSİS) = Tobacco Addiction Psychological Support Programme) based on mindfulness psychological intervention with a web-based, online platform-supported application for male and female individuals over the age of 18 with tobacco use. The TÜBSİS Programme, which is an individual intervention, was applied to male and female tobacco users at a university via a web platform.

Method: In this randomised controlled study, data collection from the participants in the intervention group was carried out through the web-based platform of the TÜBSİS Programme. Data collection from the participants in the control group was carried out via Google Forms and Google E-mail (Gmail). The participants were asked questions including the intervention variables three times in total, at the beginning, after two weeks and after four weeks. The participants in the intervention and control groups were asked about sociodemographic characteristics and tobacco use characteristics at baseline. Health Action Process Approach (HAPA) Model Change Question Form, Warwick Edinburgh Mental Well-Being Scale, Fagerström Nicotine Dependence Test and Informed Consent Form were applied to both groups at the beginning, in the middle and at the end of the intervention study. Intervention Variable '4-week TÜBSİS Tobacco Addiction Psychoeducation Programme' and 'Control Variables' Sociodemographic Characteristics (Age, Gender, Education level, Student status (being a student or not and level of education), Regular employment status (present/absent), Marital status, Having children, Perceived monthly income level, Father's education level, Living environment), Tobacco Use Characteristics (Age at the time of first smoking attempt, Past (pre-survey) smoking cessation attempt and number of attempts). The primary outcomes evaluated completed-8 modules of follow-up during the TÜBSİS Programme are as follows: 'Stage of change according to the HAPA Model (pre-intender stage, intender stage, actor stage)', "7-day point prevalence smoking cessation attempt (i.e. not having smoked a puff of cigarette in the last 7 days)", "Daily cigarette consumption amount (number of cigarettes smoked in a typical day for daily smokers, number of days smoked in a month and number of cigarettes smoked in a typical smoking day for occasional smokers)". Secondary outcomes were 'Increase in Warwick Edinburgh Mental Well-being Scale score' and 'Increase in Fagerström Nicotine Dependence Test score'. All statistical analyses were performed using SPSS version 25 software.

Keywords: tobacco use, mindfulness, web-based psychoeducation, Health Action Process Approach

DETAILED DESCRIPTION:
Tobacco addiction is not only a behavioral challenge but also a neurobiological and psychosocial condition requiring tailored interventions beyond simple awareness efforts. Digital interventions-particularly those grounded in psychological theory and structured learning-have shown growing promise in addressing addictive behaviors in accessible and scalable formats.

The TÜBSİS Programme was developed as a structured psychoeducational tool incorporating principles of mindfulness and behavior change, aiming to strengthen psychological resources such as self-regulation, motivation, and resilience in tobacco users. While the program was digitally delivered, its design emphasized individual reflection, staged goal-setting, and emotional regulation skills to facilitate both cognitive and behavioral disengagement from tobacco use.

Each module of TÜBSİS was designed to align with the core constructs of the Health Action Process Approach (HAPA), such as risk perception, action self-efficacy, planning, and maintenance self-efficacy. Participants were guided through these constructs in a phased format, enabling a personalized change trajectory based on their psychological readiness and behavioral intentions.

In addition to the behavior change model, mindfulness strategies were embedded throughout the program, including attentional control exercises, present-moment awareness tasks, and cognitive reframing components. These were introduced progressively across modules to avoid cognitive overload and to allow integration into daily life routines.

Assessments used in this study were not only intended to track behavioral change but also to understand the interplay between tobacco dependence and psychological well-being. The Warwick Edinburgh Mental Well-Being Scale and the Fagerström Test provided quantitative indices of mental health status and addiction severity, allowing for multidimensional evaluation.

Given the asynchronous format, the study emphasized user engagement and retention. Platform analytics and module completion rates were monitored to interpret efficacy within the context of adherence.

ELIGIBILITY:
Inclusion criteria for the participants in the study:

* 18 years of age or older
* Used tobacco at least once a week for the last one month
* Being literate in Turkish language
* Be a student of Ege University or have graduated within the last three months

Exclusion criteria for the participants in the study:

* Currently taking any smoking cessation intervention or medical treatment
* Not having given the mid-test or post-test measurement within 3 months from the time of the pre-test in the TÜBSİS Program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Stage of Change Based on the Health Action Process Approach | Up to 12 weeks
  Participants' readiness to quit smoking is classified into one of three stages defined by HAPA model: pre-intender, intender, or actor. Stage classification is based on responses to HAPA Questionnaire.
  Unit of Measure: Stage (categorical: pre-intender, intender, actor)
7-day point prevalence smoking cessation attempt (i.e. not having smoked a puff of cigarette in the last 7 days) | Up to 12 weeks
  Defined as complete self-reported abstinence from smoking-not even a single puff-for at least the 7 days preceding the follow-up assessment.
  Unit of Measure: Percentage of participants (%)
Daily cigarette consumption amount | Up to 12 weeks
  Daily smokers will report the average number of cigarettes smoked per day. Occasional smokers will report the number of smoking days per month and the average number of cigarettes per smoking day.
  Unit of Measure: Number of cigarettes per day or per month

SECONDARY OUTCOMES:
Increase in Warwick Edinburgh Mental Well-being Scale score (Warwick-Edinburgh Mental Well-Being Scale - Short Form) | Up to 12 weeks
  Participants' mental well-being is assessed using the validated short-form Warwick-Edinburgh Mental Well-Being Scale (WEMWBS-KF). Change in total score from baseline to 12 weeks is evaluated.
  Unit of Measure: Scale score (min. score: 7 points - max. score: 35 points)
Increase in Fagerström Nicotine Dependence Test score (Fagerström Test for Nicotine Dependence) | Up to 12 weeks
  Participants' level of nicotine dependence is assessed using the Fagerström Test for Nicotine Dependence (FNBT). Change in total score from baseline to 12 weeks is evaluated.
  Unit of Measure: Scale score (min. score: 0 point - max. score: 10 points)

CONTACTS AND LOCATIONS:
Overall Officials: Gorkem YARARBAS, Prof. Dr., Principal Investigator — Ege University, Institute on Drug Abuse, Toxicology and Pharmaceutical Science, Department of Drug Abuse; Hur HASSOY, Prof. Dr., Principal Investigator — Ege University, Faculty of Medicine, Department of Public Health
Locations (1):
- Ege University Institute on Drug Abuse, Toxicology and Pharmaceutical Science, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schaub, M.P. (2023). Nikotinabhängigkeit. In: Ebert, D.D., Baumeister, H. (eds) Digitale Gesundheitsinterventionen. Springer, Berlin, Heidelberg.
- [Background] Cetin MB, Sezgin Y, Akinci S, Bakirarar B. Evaluating the Impacts of Some Etiologically Relevant Factors on Excessive Gingival Display. Int J Periodontics Restorative Dent. 2021 May/June;41(3):e73-e80. doi: 10.11607/prd.5475. Epub 2021 Apr 5. PMID 33819318
- [Background] Spears CA, Abroms LC, Glass CR, Hedeker D, Eriksen MP, Cottrell-Daniels C, Tran BQ, Wetter DW. Mindfulness-Based Smoking Cessation Enhanced With Mobile Technology (iQuit Mindfully): Pilot Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Jun 24;7(6):e13059. doi: 10.2196/13059. PMID 31237242
- [Background] van Emmerik AAP, Berings F, Lancee J. Efficacy of a Mindfulness-Based Mobile Application: a Randomized Waiting-List Controlled Trial. Mindfulness (N Y). 2018;9(1):187-198. doi: 10.1007/s12671-017-0761-7. Epub 2017 Jun 21. PMID 29387266
- [Background] Thornton L, Quinn C, Birrell L, Guillaumier A, Shaw B, Forbes E, Deady M, Kay-Lambkin F. Free smoking cessation mobile apps available in Australia: a quality review and content analysis. Aust N Z J Public Health. 2017 Dec;41(6):625-630. doi: 10.1111/1753-6405.12688. Epub 2017 Jul 27. PMID 28749591
- [Background] Oikonomou MT, Arvanitis M, Sokolove RL. Mindfulness training for smoking cessation: A meta-analysis of randomized-controlled trials. J Health Psychol. 2017 Dec;22(14):1841-1850. doi: 10.1177/1359105316637667. Epub 2016 Apr 4. PMID 27044630
- [Background] Firat M, Demir Gokmen B, Karakurt P. An investigation of smoking habits and mental well-being in healthcare personnel during COVID-19. Perspect Psychiatr Care. 2022 Jan;58(1):108-113. doi: 10.1111/ppc.12819. Epub 2021 Apr 30. PMID 33931894
- [Background] Legleye S, Bricard D, Khlat M. Roles of parental smoking and family structure for the explanation of socio-economic inequalities in adolescent smoking. Addiction. 2023 Jan;118(1):149-159. doi: 10.1111/add.16026. Epub 2022 Aug 26. PMID 35971293
- [Background] Haug S, Paz Castro R, Kowatsch T, Filler A, Dey M, Schaub MP. Efficacy of a web- and text messaging-based intervention to reduce problem drinking in adolescents: Results of a cluster-randomized controlled trial. J Consult Clin Psychol. 2017 Feb;85(2):147-159. doi: 10.1037/ccp0000138. Epub 2016 Sep 8. PMID 27606700
- [Background] Haug S, Schaub MP, Venzin V, Meyer C, John U. Efficacy of a text message-based smoking cessation intervention for young people: a cluster randomized controlled trial. J Med Internet Res. 2013 Aug 16;15(8):e171. doi: 10.2196/jmir.2636. PMID 23956024
- [Background] Durmaz S, Ergin I, Durusoy R, Hassoy H, Caliskan A, Okyay P. WhatsApp embedded in routine service delivery for smoking cessation: effects on abstinence rates in a randomized controlled study. BMC Public Health. 2019 Apr 8;19(1):387. doi: 10.1186/s12889-019-6727-z. PMID 30961557
- [Background] Bandura, A. (1969). Social-learning theory of identificatory processes. In D. A. Goslin (Ed.), Handbook of socialization theory and research (pp. 213-262). Chicago, IL: Rand McNally.